CLINICAL TRIAL: NCT06383598
Title: PD-L1 Specific 68Ga-THP-PD-L1-3 Probe for PET Imaging in Solid Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hua Zhu (Other)
Responsible Party: Sponsor-Investigator, Hua Zhu, Principal Investigator, Peking University Cancer Hospital & Institute
Organization: Peking University Cancer Hospital & Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022KT74-ZY01
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 68Ga-THP-PD-L1-3 (Experimental): All study participants will be allocated to this arm (single-arm study).Study participants will undergo 68Ga-THP-PD-L1-3 PET/CT scans (At the investigator's discretion, a total of no more than 0.5 mg of non-radiolabeled precursor may be considered for injection. To reduce liver and bone marrow uptake). After resting for 40 minutes or 1 hour, participants underwent United Imaging Healthcare total-body PET/CT for whole body scans or a Siemens Biograph m-CT flow PET/CT from the top of the head to the upper third of the thighs.
  Interventions: Drug: 18F-FDG

INTERVENTIONS:
Drug: 18F-FDG — All study participants will undergo one 18F-FDG PET/CT scan.

SUMMARY:
The objective of the study is to constrcut a noninvasive approach 68Ga-THP-PD-L1-3 PET/CT to detect the PD-L1 expression of tumor lesions in patients with solid tumors and to identify patients benefiting from anti-PD-L1 treatment.

DETAILED DESCRIPTION:
Analysis plan: 1. recruit 10 participants to analyze preliminary pharmacokinetic/first-in-human dose (FIH), major organ distribution and tumor uptake information via whole-body PET/CT imaging; 2. recruit 20-30 participants to analyze in vivo safety and tumor targeting information; and 3. recruit all participants for a final summary.

ELIGIBILITY:
Inclusion Criteria:

1. Aged >18 years old; ECOG 0 or 1;
2. Patients with solid tumorsin or suspected tumor lesions;
3. life expectancy >=12 weeks.

Exclusion Criteria:

1. Significant hepatic or renal dysfunction;
2. Is pregnant or ready to pregnant;
3. Cannot keep their states for half an hour;
4. Refusal to join the clinical study;
5. Suffering from claustrophobia or other mental diseases;
6. Any other situation that researchers think it is not suitable to participate in the experiment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value（SUV） | 2 years
  The uptake of the tracer （68Ga-THP-PD-L1-3) in solid tumor lesions or suspected tumor lesions by measuring SUV on PET/CT.

CONTACTS AND LOCATIONS:
Overall Officials: Hua Zhu, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China